CLINICAL TRIAL: NCT07226037
Title: Development of Systems and Education for Cervical Cancer Prevention (DOSE-CC)
Acronym: DOSE-CC
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: H-46139; R01CA299475 (NIH)
Record Dates: First submitted 2025-11-06; First posted 2025-11-10 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Cervical Cancer Screening; Cervical Cancer
Keywords: DOSE-CC; cervical cancer; prevention
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Intervention Model Description: Step wedge randomized trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DOSE-CC Intervention: Educational Sessions (Experimental): The primary goals of the DOSE-CC intervention are to 1) use education and training to increase clinician motivation to provide guideline-concordant screening and follow-up and reduce missed opportunities, and 2) support systems changes to improve screening and follow-up processes. Repeated contacts with clinicians will be used to reinforce learned concepts and motivate participants to achieve their goals. The first two sessions will follow a standardized curriculum, while the last three sessions will include development and implementation of tailored activities designed to address systems barriers and meet individual practice needs.
  Interventions: Behavioral: DOSE-CC Intervention: Educational Sessions

INTERVENTIONS:
Behavioral: DOSE-CC Intervention: Educational Sessions — Session 1: Introduction to the project, and feedback/discussion around clinic screening rates.
  Session 2: Education on cervical cancer, impact of screening on cancer prevention and health equity, different methods of screening, and recent updates to screening and follow-up guidelines.
  Session 3: Action plan development. Sessions 4 and 5: Quality improvement through plan-do-study-act cycles and assessment of the success of the action plan.

SUMMARY:
Cervical cancer disproportionately impacts those who have not accessed screening or follow-up. Universal screening has the potential to decrease the overall burden of cervical cancer. However, more than half of the individuals who develop cervical cancer have not been screened in more than 5 years, and 20% did not follow-up after an abnormal result.

To address this problem, the investigators will adapt and test an intervention to improve cervical screening and follow-up in three different settings: Northeastern US urban inner city (Boston), Southeastern US suburban (Florida), and remote west, rural (Hawaii). Our research group previously developed a successful intervention to improve primary cervical cancer prevention, which will be adapted for cervical cancer screening. The intervention combines education and quality improvement methods using a mechanism called Performance Improvement Continuing Medical Education. This type of intervention is attractive to clinicians because they are able to improve their cancer prevention practices while fulfilling requirements for maintaining board certification.

When applied to primary prevention, the intervention improved rates by over 10 percentage points, and gains continued for over 4 years after the intervention concluded. The goal of the proposed research is to adapt the intervention to cervical cancer screening, and to evaluate its effectiveness in improving cervical cancer screening and follow-up after abnormal results.

The proposed intervention represents an innovative and scalable model for promoting cancer prevention and screening activities by clinicians. Unlike programs that increase administrative burdens on busy clinicians, the proposed intervention allows clinicians to improve cancer prevention practices while simultaneously fulfilling requirements to maintain their board certification and improving the quality of cancer prevention care. It therefore has great potential for widespread dissemination.

DETAILED DESCRIPTION:
The research will specifically address the following objectives.

First, the investigators' successful primary prevention intervention will be adapted to address cervical cancer screening (DOSE-CC [Development of Systems and Education for Cervical Cancer Prevention]). Key stakeholders will be interviewed to explore facilitators and barriers to screening and follow-up at the patient, clinician, and healthcare setting levels and use these findings and Advisory Board input to develop the DOSE-CC intervention.

Second, the investigators will validate DOSE-CC using a Hybrid Type 1 effectiveness-implementation, stepped wedge randomized controlled trial design of the 6-month intervention, reaching over 40,000 patients.

Third, guided by the RE-AIM QuEST (Reach, Effectiveness, Adoption, Implementation Qualitative Evaluation for Systemic Translation) framework, the investigators will conduct semi-structured interviews of key stakeholders to examine intervention reach, adoption, implementation, maintenance and sustainability, and barriers and facilitators of intervention success.

ELIGIBILITY:
Inclusion Criteria:

* Active patients (defined as having a primary care provider assigned at the clinical site and with an appointment in the past 18 months)
* Eligible for cervical cancer screening (e.g., has a cervix and not up to date with screening)

Exclusion Criteria:

* None

Ages: 21 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80000 (Estimated)
Dates: Start 2027-05 (Estimated); Primary Completion 2029-05 (Estimated); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants who receive cervical cancer screening | 1-5 years, depending on prior test and result
  Defined as a cervical cytology (Pap test) and/or HPV test for those who are due

SECONDARY OUTCOMES:
Number of participants with diagnostic resolution among those with abnormal screening results per 2019 ASCCP guidelines | 18 months
  (e.g., receipt of colposcopy, treatment, additional follow-up testing)

CONTACTS AND LOCATIONS:
Overall Officials: Lunze Karsten, MD, MPH, Principal Investigator — Boston Medical Center, General Internal Medicine

IPD SHARING:
Plan to Share IPD: No